CLINICAL TRIAL: NCT04123002
Title: Effect of Miswak on P.Gingivalis
Brief Title: Effect of Miswak Chewing Sticks on Periodontal Pathogens and Its Impact on the Progression of Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud Bin Abdulaziz University for Health Sciences (Other)
Collaborators: Kuwait University (Other)
Responsible Party: Principal Investigator, Dr Jagan K Baskaradoss, Assistant Professor, Kuwait University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: FOD6
Record Dates: First submitted 2019-10-03; First posted 2019-10-10 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Gingivitis
Keywords: P.gingivalis; Miswak
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Study participants would be divided into 2 groups. Group A would received tooth brush and paste and Group B would receive Miswak chewing stick along with tooth brush and paste. They would be instructed to use the assigned oral hygiene aid for a week. Then the groups would cross-over and continue for 1 week. Plaque and gingival measures would be taken at baseline, end of week 1 and end of week 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Miswak chewing sticks would be provided to the participants and they would be explained the method of use
  Interventions: Other: Miswak chewing sticks
- Comparison group (No Intervention): They would use only tooth brush and paste

INTERVENTIONS:
Other: Miswak chewing sticks — Chewing stick are routinely used by this population
  Arms: Interventional group

SUMMARY:
A cross over randomized clinical trial Group A- Tooth Brush and Paste only Group B- Tooth Brush and Paste and Miswak chewing sticks

DETAILED DESCRIPTION:
The study design would be a cross over randomized clinical trial. The study sample would be selected from the regular dental patients visiting the Faculty of Dentistry, Kuwait University, Kuwait. The subjects of our study are patients with >24 teeth who are physically/mentally healthy and those who were diagnosed with gingivitis. There will be an initial screening of the subjects, where patients would be briefed on the study components and informed consent would be obtained from those who are willing to participate in this study. The study subjects would be randomly divided into two groups; Group 1 subjects would be instructed to brush their teeth two times per day, in the morning and in the evening before going to the bed, and to refrain from using a miswak during this period. Group 2 subjects would receive the same instructions as Group 1 subject, but, in addition, they would also be instructed to use miswak chewing sticks two times a day. All the participants would then be given instructions on how to use miswak and toothbrush by the investigators. A sample size of 20 was considered sufficient to conduct this study. The socio-demographic details of the study participants would be obtained from the electronic dental records. Plaque index and gingival bleeding index would be taken at baseline and on day 14. Plaque samples would be collected at baseline - before and after the intervention (tooth brushing/miswak), day 3, day 7 and day 14. The oral plaque samples would be sent for PCR analysis.

Randomized assignment of the subjects regarding the order of miswak and toothbrush would be carried out, by a random binary outcome of a dice, even or odd numbers. Group 1 subjects would be given a new toothbrush (regular, straight handled Oral-B toothbrush). Group 2 subjects would also be given a new toothbrush (regular, straight handled Oral-B toothbrush) as well as 14 fresh sticks of miswak (20 cm in length and 7mm in width) to be used daily. Then the groups would be crossed over.

Sample collection procedure and Purification of Microbes Subgingival and supragingival plaques samples would be collected using a sterile universal curette. Subgingival plaque samples would be collected from the deepest periodontal pocket. The sampling area would be isolated from saliva and gently dried with air. The point would be then immersed in 0.5 ml sterile distilled water in Eppendorf tubes (epTIPS Standard, Eppendorf AG, Hamburg, Germany). The collected samples would be then sent to the Microbiology Laboratory, Faculty of Dentistry, Kuwait University and PCR analysis would be conducted to identify the strains.

ELIGIBILITY:
Inclusion Criteria:

* The subjects of our study are patients with >24 teeth who are physically/mentally healthy
* Those who were diagnosed with gingivitis. There will be an initial screening of the subjects, where patients would be briefed on the study components and informed consent would be obtained from those who are willing to participate in this study

Exclusion Criteria:

* Patients on antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
The gingival health of index teeth as measured using a standardized index | 2 weeks
  Gingival health would be measured using Loe and Silness gingival index

CONTACTS AND LOCATIONS:
Locations (2):
- Kuwait (2):
  - Jagan K Baskaradoss, Kuwait City
  - Kuwait University, faculty of dentistry, Kuwait City